CLINICAL TRIAL: NCT04282044
Title: A Phase 1 Study of the Safety and Efficacy of CRX100 as Monotherapy and in Combination With Pembrolizumab in Advanced Solid Malignancies
Brief Title: Study of CRX100 as Monotherapy and in Combination With Pembrolizumab in Patients With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioEclipse Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRX100-001
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor, Adult; Triple Negative Breast Cancer; Colorectal Cancer; Hepatocellular Carcinoma; Osteosarcoma; Epithelial Ovarian Cancer; Gastric Cancer; Non-small Cell Lung Cancer; Malignant Melanoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Colorectal Neoplasms; Carcinoma, Hepatocellular; Osteosarcoma; Carcinoma, Ovarian Epithelial; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy Dose-Escalation Cohorts (Experimental): Prior to the current amendment, no DLTs were observed at Dose Levels 1-5. Starting with the current protocol amendment, dosing decisions in monotherapy cohorts will utilize a 3+3 design for Dose Level 6. CRX100 infusion will occur every nine weeks (+/- 7 days). Subjects will receive up to a maximum of four infusions of CRX100 unless it is determined by the treating physician and the sponsor that it is in the best interest of the subjects to receive additional doses of CRX100 beyond four doses. A minimum of three DLT-evaluable subjects will be doses at Dose Level 6 and expanded to six subjects if determined necessary based on DLT incidence using the 3+3 design, and discussion with SRC and Sponsor.
  Interventions: Biological: CRX100 suspension for infusion; Combination Product: Fludarabine; Combination Product: Cyclophosphamide
- Combination Therapy Cohorts (Experimental): Subjects with relasped or refractory solid tumors, as defined in the inclusion criteria, will be enrolled to evaluate the safety and anti-tumor activity of CRX100 in combination with Pembrolizumab in patients with advanced solid malignancies. The dose of CRX100 used will be determined from the monotherapy cohorts.
  CRX100 infusion will occur every nine weeks (+/- 7 days). Subjects will receive up to a maximum of four doses of CRX100 unless it is determined by the treating physician and the sponsor that it is in the best interest of the subjects to receive additional doses of CRX100 beyond four doses.
  Pembrolizumab will be administered at 200mg IV every three weeks (Q3W) per the approved label.
  Interventions: Biological: CRX100 suspension for infusion; Combination Product: Fludarabine; Combination Product: Cyclophosphamide

INTERVENTIONS:
Biological: CRX100 suspension for infusion — A fixed dose of CIK cells combined with the specified dose of CDSR.
Combination Product: Fludarabine — 25mg/m IV (five doses given from Day -7 until Day -3)
Combination Product: Cyclophosphamide — 60mg/kg intravenous (IV) (two doses given on Day -7 and -6)

SUMMARY:
This clinical study is an open-label, Phase 1, dose-escalation study to determine the safety, tolerability, and efficacy of the drug product produced by Administering CRX100 alone and in combination with Pembrolizumab in advanced solid malignancies. Patients will be screened and evaluated to determine whether or not they meet stated inclusion criteria. Enrolled subjects will undergo leukapheresis to enable the ex vivo generation of CRX100. Patients with non-small cell lung cancer (NSCLC), ovarian cancer, colorectal cancer, hepatocellular carcinoma (HCC), malignant melanoma (excluding uveal melanoma), gastric cancer, triple negative breast cancer, and osteosarcoma.

The study will start with monotherapy dose escalation followed by combination cohorts.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be enrolled in this study:

1. Age ≥18 years at the time of consent.
2. Written informed consent in accordance with national, local, and institutional guidelines obtained prior to any study procedures. (Screening assessments performed prior to informed consent but within the 28-day screening window are acceptable for inclusion purposes).
3. Subjects must have histologically confirmed diagnosis of one of the following tumors: triple negative adenocarcinoma of the breast (human epidermal growth factor receptor 2 negative, estrogen receptor negative and progesterone receptor negative [HER2-/ER-/PR-]), adenocarcinoma of the colon or rectum, hepatocellular carcinoma (HCC), osteosarcoma, epithelial ovarian cancer, malignant melanoma, non-small cell lung cancer (NSCLC), or gastric cancer. Documentation of the diagnosis with the original pathology report, or a recent biopsy, is required.
4. Subjects must have relapsed disease or refractory disease. Subjects must have received, completed, or become intolerant of prior standard of care therapies or are not expected to derive any clinical benefit from standard of care therapies.
5. Subjects with Ovarian cancer must have received at least one prior standard of care for their relapsed or refractory disease, which must include a platinum-based regimen.
6. Subjects agree to provide fresh tumor tissue that has not been previously irradiated. If biopsy procedure is not safe to perform, then archival tumor tissue (20 slides or a tissue block) can be submitted.
7. Subjects must have iRECIST evaluable disease using computed tomography (CT) or magnetic resonance imaging (MRI) with IV contrast, with at least one measurable target lesion.
8. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
9. Subjects are expected to have a life expectancy of at least 12 weeks from the time of enrollment.
10. Adequate hematologic function at the time of screening, defined as: absolute lymphocyte count (ALC) >500 cells/mm3, absolute neutrophil count (ANC) >750 cells/mm3, hemoglobin >8 g/dL, and platelet count >50,000 cells/mm3. For subjects enrolling into the LDC cohorts, the criteria are defined as: ALC>500 cells/mm3, ANC>1000 cells/mm3, hemoglobin>8g/dL, and platelet count>100,000 cells/mm3.

    a. Hemoglobin and platelet count thresholds must be achievable without transfusion of red blood cells or platelets, or use of growth factors administered within two weeks.
11. Adequate organ function, defined as:

    1. Renal function: serum creatinine <1.5x institutional upper limit of normal (ULN) or calculated creatinine clearance >50 mL/min.
    2. Adequate hepatic function: total bilirubin ≤1.5x institutional ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5x institutional ULN, unless liver metastases are present, in which case it must be ≤5x ULN; International Normalized Ratio (INR) ≤1.5. For subjects with HCC, adequate hepatic function is defined as: total bilirubin ≤3x institutional upper limit of normal, AST/ALT ≤5x institutional ULN, INR ≤1.7, Child-Turcotte-Pugh score <8.
12. Women of childbearing potential (defined as all subjects physiologically capable of becoming pregnant) must have negative serum ß-human chorionic gonadotropin (hCG) or urine pregnancy test.
13. Women of childbearing potential must agree to use highly effective methods of contraception throughout the study and for six months after the last dose of CRX100.
14. Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method throughout the study and for six months after the last dose of CRX100.
15. Subjects must be willing and able to comply with all study procedures, requirements, and follow-up examinations.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participation in this study:

1. Subjects with new or progressive brain metastasis. Subjects with treated brain metastases are eligible if there is no evidence of progression for at least four weeks after central nervous system-directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period.
2. Subjects who received any chemotherapy or immunotherapies (non-cell-based therapies) or oncolytic virus therapy, radiotherapy, radiosurgery or investigational agents within three weeks of enrollment.
3. Subjects who still are experiencing Grade 2 or higher AEs from prior therapies such as surgery, radiation therapy and systemic anti-cancer therapies unless approved by sponsor.
4. Subjects who received any type of cell-based therapies within the last 12 weeks from the planned apheresis date.
5. Subjects experiencing any active infections (bacterial, viral, or fungal) for which systemic antimicrobials are required. Subjects who need prophylactic anti-viral agents that can inhibit the replication of VACV will be excluded from participating.
6. Subjects must not have history of active or symptomatic autoimmune disease or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, other symptomatic autoimmune disease, documented history of autoimmune disease or syndrome requiring systemic treatment in the past two years (i.e., with use of disease modifying agents, steroids or immunosuppressive agents) Exceptions are permitted for vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition requiring only hormone replacement, psoriasis not requiring systemic treatment, conditions not expected to recur in the absence of an external trigger or other conditions approved by the medical monitor.
7. Have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days prior to apheresis, and within 14 days prior to infusion. Inhaled, intramuscular injection, or topical steroids and adrenal replacement doses (≤10 mg daily prednisone equivalents) are permitted. Stable doses of steroids are permitted for subjects with pre-treated brain metastases. Short-term (<48 hr) steroid pretreatment for contrast allergy for imaging is permitted.
8. Known human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C, life-threatening illnesses unrelated to cancer, or any serious medical or psychiatric illness that could, in the Investigator's opinion, interfere with participation in this study.
9. Pregnant or nursing an infant (subject or household contacts).
10. Clinically significant immunodeficiency (e.g., due to underlying illness and/or medication) in a subject or household contacts.
11. Have any underlying medical condition (including, but not limited to, ongoing or active infection requiring treatment, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia), psychiatric condition that, in the opinion of the Investigator, would compromise study administration as per protocol or compromise the assessment of AEs.
12. Have a history of another invasive malignancy, except for the following circumstance: individuals with a history of invasive malignancy are eligible if they have been disease free and off treatment for at least two years or are deemed by the Investigator to be at low risk for recurrence of that malignancy; individuals with the following cancers are eligible if diagnosed and treated: carcinoma in situ of the breast, oral cavity, or cervix, localized prostate cancer, or basal cell or squamous cell carcinoma of the skin. When enrolling a subject with another malignancy, the Investigator must discuss the subject with the Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment-emergent Adverse Events and Dose Limiting Toxicities | 28 days following dose administration for each dosed subject.
  The Primary Outcome Measure will be based on the frequency of treatment-emergent Adverse Events and Dose Limiting Toxicities during and after the administration of investigational drug in monotherapy and investigational drug with combination therapy.
Determine the maximum tolerated dose (MTD), maximum feasible dose (MFD) or optimal biological dose (OBD) and determine recommended Phase 1b/Phase 2a dose level. | 28 days following dose administration for each dosed subject.
  Review of safety review committee following subject treatment to review any AEs, SAEs, or DLTs

SECONDARY OUTCOMES:
Biodistribution of CRX100 based on subject's viral load as assessed through a viral shedding assay. | 28 days following dose administration for each dosed subject.
  To characterize the biodistribution of CRX100 based on each subject's viral load as assessed through a viral shedding assay, following a single dose of investigational product.
Immune response to investigational drug based on subject's levels of neutralizing antibodies. | 28 days following dose administration for each dosed subject.
  Levels of neutralizing vvDD antibodies will be summarized by dose level and time point following a single dose of investigational product.
Early anti-tumor activity of investigational drug based on iRECIST criteria | 6 months after dose administration for each dosed subject.
  Summarized based on best response observed using RECIST classification of response. Overall response and frequencies of each level of response.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Dorigo, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Stanford University, Stanford, California